CLINICAL TRIAL: NCT06557655
Title: The Effect of Caffeinate Chewing Gum on Ice Hockey Performance After Partial Sleep Deprivation: a Double-blind Crossover Trial
Brief Title: Caffeinate Chewing Gum on Ice Hockey Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Chih-Hui Chiu, Professor, National Taiwan Sport University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 113-4
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Caffeine; Placebo
Keywords: exercise performance; fatigue index

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The order of participants was determined through the use of computerized randomization software
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caffeine gum (Experimental): 15 minutes before exercise
  Interventions: Dietary Supplement: caffeinate chewing gum
- placebo (Placebo Comparator): 15 minutes before exercise
  Interventions: Dietary Supplement: caffeinate chewing gum

INTERVENTIONS:
Dietary Supplement: caffeinate chewing gum — participants either chewed caffeinated gum (CAF) containing 3 mg/kg caffeine or a caffeine-free placebo gum (PLA) for 10 minutes prior to undertaking a series of tests on-ice and off-ice.
  Other Names: plocabo gum

SUMMARY:
The purpose of this study was to examine the impact of caffeinated chewing gum on the physical performance of elite ice hockey players in a partial sleep deprivation state.

DETAILED DESCRIPTION:
This study used a randomisation crossover design with a single-blind, double-blind experimental design. The participants were randomly assigned to either a caffeinated chewing gum trial (CAF) or a placebo trial (PL).

ELIGIBILITY:
Inclusion Criteria:

* 1. 6 years of professional ice hockey training,
* 2. 6 months of continuous training,
* 3. 3 months of recovery from sports injuries such as strains and sprains

Exclusion Criteria:

* 1. non-specialised ice hockey player.
* 2. has not trained regularly for the past 6 months.
* 3. has recovered from an athletic injury.
* 4. have been recovering from a sports injury for less than 3 months, or have epilepsy, hypertension, hyperlipidemia, heart disease, arthritis, osteoporosis, brain injury, or a history of caffeine allergy.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only health male players
Enrollment: 14 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
counter-movement jump | 15 minutes after intervention
  jump height

SECONDARY OUTCOMES:
35-metre sprint | 15 minutes after intervention
  complete time (seconds)

CONTACTS AND LOCATIONS:
Overall Officials: ChihHui Chiu, PhD, Study Director — National Taiwan University of Sport
Locations (1):
- National Taiwan University of Sport, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
No IPD plan available

DOCUMENTS (1):
  • Study Protocol (2024-08-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT06557655/Prot_000.pdf